CLINICAL TRIAL: NCT01591824
Title: Effectiveness of Resonant Oscillation, According to the Pold Concept in Chronic Nonspecific Low Back Pain
Brief Title: Study of Effectiveness of Pold in Chronic Nonspecific Low Back Pain
Acronym: Pold-LBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omphis Foundation (Other)
Responsible Party: Principal Investigator, JUAN V. LOPEZ DIAZ, Degree in physiotherapy kinesiology and physiatry, Omphis Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pold-LBP
Record Dates: First submitted 2012-05-01; First posted 2012-05-04 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Mechanical Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Functional Laterality

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- POLD TREATMENT (Experimental): Patients who applies the treatment of resonant oscillation according to the Pold Concept
  Interventions: Other: Resonant oscillation
- CONVENCIONAL: column exercise group (Active Comparator): Patients who applied the conventional treatment of hospital
  Interventions: Other: column exercise group

INTERVENTIONS:
Other: Resonant oscillation — Resonant sustained oscillations are applied in the following areas
  * general column.
  * lumbar muscles, and paraspinal muscles,
  * sacral decompression oscillatory
  * Opening by lateral vertebral lumbar rhythmic swing.
  * Balancing and pelvic decompression
  * Swing-lumbar vertebral rotation.
  Other Names: oscillatory movement
  Arms: POLD TREATMENT
Other: column exercise group — * paraspinal muscle stretching exercises
  * postural correction
  * mobilization exercises thoracic and lumbar
  * Motor control exercises
  Other Names: motor control
  Arms: CONVENCIONAL: column exercise group

SUMMARY:
Through this research is to conduct a pilot clinical trial in the treatment of chronic nonspecific low back pain (degenerative and mechanical), by comparing two groups, one that will apply a technique of physiotherapy by passive movement of the column with oscillations in axial rotation at a frequency of 1.5 to 2 cps (resonance) of low amplitude (called "Pold Concept"), another group that applies the standard protocol of treatment for this condition, as used in the hospital where performed the study.

It will compare the levels of efficiency and effectiveness of each treatment and the comparison between them. This will measure the perception of pain intensity and disability.

DETAILED DESCRIPTION:
Type of study:

This is an analytical study, the experimental group clinical trial type, controlled, randomized with complete randomization and single blind.

Two groups, the study to which the POLD treatment shall apply, and the control group with conventional treatment will be formed by complete randomization system as they arrive for consultation, with a total of 50 patients or more if they were needed for each group have a minimum of 25 having offset dropouts. The number of 25 patients per group is determined considering accepting an alpha risk of 0.05 and a beta risk of 0.20 in a bilateral contrast, are required at least 21 subjects in each group to detect a minimum difference of 15 percentage points between the two groups, therefore two groups of 25 assuming a standard deviation of 15 points and a loss rate of 0% tracking form.

We will study both the effectiveness and efficiency individually and comparatively between groups.

* Study population:

  1. The sample was selected from patients attending the clinic with back pain and after medical diagnosis are referred to the physiotherapist report of diagnosis, prescribing physical therapy and who meet the criteria for inclusion and not exclusion .
  2. A total of 25 patients in the experimental group and 25 for the standard treatment group are selected.
  3. If losses to the sample will be replaced by others to maintain proportions.
* The selection of groups:

RANDOM will be used , he formed the experimental group and control directing patients overall are being incorporated randomly according to the study :

1. Group A ( study ) will apply the technique with an identical protocol POLD them all.

2. Group B (conventional control) was applied average conventional treatment of different physiotherapy centers of reference.

* Study variables to collect:

  1. Subjective assessment of pain intensity using VAS, visual analog pain. ,
  2. Evolution of disability by Oswestry test.
  3. SF-12 on health.
* Statistical analysis:

Computer analysis using "SPSS" 13.0 ® processed program. The study will be processed as follows:

First, an initial analysis was performed to verify that there were no significant differences between groups in baseline values of the dependent variables by Student's t test for independent samples.

Second : For each dependent variable variance analysis is applied using a general linear model with 2x10 between subjects factor we call variable " Treatment " with two categories 1, 2 (experimental group = 1, conventional group = 2 ) and a temporal within-subjects factor we call "SHOOT" ( 10 sessions) .

Third: We analyze to what treatment session the differences between the two groups appear by Student's t test for independent data after the first session

Fourth, the interactions are studied by comparing the two groups after the first, fifth and 10th session using a Student t test for independent data and comparing the results of each group between 1st and 5th session and between 1st and 10th session with a Student t for paired data.

• Ethical Issues: During the study of national and international guidelines (code of ethics, Declaration of Helsinki) will continue, likewise the legal regulations on data privacy (Law 15 /1999 of 13 December on the Protection of Personal Data)

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis instrumental prior to treatment to rule out pathologies pollutants, neurological or structural malformations.
* No previous trauma.
* Age between 25 and 65.
* With similar clinical characteristics to have a homogenous group:

  * Low back pain (> 3 months) and that at the time the study began have a minimum of 3/10 on VAS scale, following the criteria established in similar studies
  * without component of neurological lower limbs irradiation

Exclusion Criteria:

* Existence of other recent traumatic structural pathologies in the lumbar region or of another type that could disturb the study.
* Existence of irradiation metameric to lower limbs
* Current tumors in the lumbar region
* Ongoing infectious disease in the lumbar area.
* Inflammatory rheumatism in the lumbar region.
* Lumbar surgery complications.
* Ongoing pregnancy.
* They have been treated with infiltrations in the last month.
* Who are following any other treatment, whether manual or physical agents or alternative or complementary therapies.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-05; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
VAS pain measurement | Participants will be followed for the duration of treatment application, an expected average of 3 weeks.
  Visual analog scale of pain measurement, with values between zero and ten where zero is total absence of pain and 10 the maximum pain imaginable by the patient, distributed in a horizontal line, without intermediate numerical or graphic references.

SECONDARY OUTCOMES:
SF-12 Health Survey | Participants will be followed for the duration of treatment application, an expected average of 3 weeks.
  The Health Questionnaire SF-12 is the adaptation made for Spain of the SF-12 Health Survey. The SF-12 is a reduced version of the SF-36 Health Questionnaire.
  This instrument provides a profile of the state of health and is one of the most widely used generic scales in the evaluation of clinical outcomes, being applicable both for the general population and for patients with a minimum age of 14 years and both in descriptive studies and in evaluation.
  It consists of 12 items from the 8 dimensions of SF-36: Physical Function (2), Social Function (1), Physical Role (2), Emotional Role (2), Mental Health (2), Vitality (1), Pain body (1), General Health (1). Response options form Likert-type scales that evaluate intensity or frequency.
  The number of response options ranges from three to six, depending on the item
Oswestry Disability Index | Participants will be followed for the duration of treatment application, an expected average of 3 weeks.
  The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel.
  Each topic category is followed by 6 statements describing different potential scenarios in the patient's life relating to the topic. The patient then checks the statement which most closely resembles their situation. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability.
  The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.

CONTACTS AND LOCATIONS:
Overall Officials: José M. Muniesa, physiatrist, Study Director — Esperanza Hospital (Barcelona)
Locations (1):
- Esperanza Hospital, Barcelona, Spain

REFERENCES:
- See also: Click here for more information about Omphis Foundation activities, Clinic, teaching and research — http://www.omphis.es